CLINICAL TRIAL: NCT01156220
Title: Investigation of Gender Specificity of the Effects of Furosemide in Healthy Female and Male Volunteers
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study was never implemented.
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IPT0901
Record Dates: First submitted 2010-07-01; First posted 2010-07-02 (Estimated); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Healthy Male and Female Volunteers
Keywords: gender, diuretics, furosemide, aminohippuric acid
MeSH Terms: conditions — Coitus | interventions — Furosemide; p-Aminohippuric Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- female (Experimental): The healthy female volunteers receive furosemide and aminohippurate sodium "PAH" as single dose randomised on day 1 or day 2.
  Interventions: Drug: Furosemide; Drug: aminohippurate sodium
- male (Experimental): The healthy male volunteers receive furosemide and aminohippurate sodium "PAH" as single dose randomised on day 1 or day 2
  Interventions: Drug: Furosemide; Drug: aminohippurate sodium

INTERVENTIONS:
Drug: Furosemide — Injection, 40 mg, single dose over 5 min
  Other Names: ATC code: C03CA01; Product name: Lasix 40 mg Injektionslösung
Drug: aminohippurate sodium — Injection, 500 mg, single dose over 5 min
  Other Names: ATC code: V04CH30,; Product name: Aminohipppurate Sodium "PAH"

SUMMARY:
In this study the gender specificity of the effects of furosemide in female and male volunteers will be investigated. The main objective is gender-specific comparison of the pharmacokinetic parameters of furosemide in relation to the effect of furosemide (urinary excretion). Secondary objectives are the gender-specific comparison of renal and systemic PAH clearance with the clearance of furosemide and the influence of various genetic polymorphisms on the variability of furosemide pharmacokinetics.

DETAILED DESCRIPTION:
In this study the gender specificity of the effects of furosemide in female and male volunteers will be investigated. The healthy volunteers receive 1. furosemide and 2. aminohippurate sodium "PAH" as single dose. The main objective is gender-specific comparison of the pharmacokinetic parameters of furosemide in relation to the effect of furosemide (urinary excretion). Secondary objectives are the gender-specific comparison of renal and systemic PAH clearance with the clearance of furosemide and the influence of various genetic polymorphisms on the variability of furosemide pharmacokinetics.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer for medical history and physical examination findings
* 18 years, <40 years
* Written informed consent is given
* No clinically relevant changes in laboratory parameters
* Inconspicuous current ECG
* taking medication under a different drug trial within the last 30 days

Exclusion Criteria:

* concomitant medication at study days or a week before
* allergies or known hypersensitivity reactions to furosemide or aminohippurate sodium
* decreased creatinine clearance by Cockcroft-Gault (<100 ml / min)
* current drug abuses
* opiate addiction within the last 10 years
* smoking within the last year
* pregnancy and 6 months postpartum, lactation
* deprivation of legal capacity
* Cooperation inability

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2012-01 (Estimated); Primary Completion 2012-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
pharmacokinetic parameter of furosemide (AUC-24) | day 1 or day 2
  Gender-specific comparison of the pharmacokinetic parameters of furosemide (AUC-24). The sample size calculation for this study was conducted with respect to the expected gender difference in the AUC24 of furosemide.
pharmacodynamic parameter of furosemide (Sodium excretion in the urine) | day 1 or day 2
  Gender-specific comparison of effect of furosemide on urinary excretion (sodium)

SECONDARY OUTCOMES:
pharmacogenetic parameters | day 1
  Influence of various genetic polymorphism (OAT1, OAT 4, OATP1B1, NKCC2, NCC, ENaC) on the variability of pharmacokinetic of furosemide
pharmacokinetic of aminohippuric acid | day 1 or day 2
  gender-specific comparison of renal and systemic PAH clearance with the clearance of furosemide
other pharmacokinetic parameter of furosemide | day 1 or day 2
  Gender-specific comparison of the other pharmacokinetic parameters of furosemide (Cmax, tmax, t½, CLoral, CLren)
other pharmacodynamic parameter of furosemide | day 1 or day 2
  Gender-specific comparison of effect of furosemide on urinary excretion (chloride, potassium, uric acid, calcium, magnesium, creatinine)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Eschenhagen, Prof.Dr.med., Study Director — Institut für Experimentelle und Klinische Pharmakologie und Toxikologie Universitätsklinikum Hamburg-Eppendorf Martinistr. 52 20246 Hamburg GERMANY; Ulrike Werner, PD Dr., Principal Investigator — Institut für Experimentelle und Klinische Pharmakologie und Toxikologie Universitätsklinikum Hamburg-Eppendorf Martinistr. 52 20246 Hamburg GERMANY
Locations (1):
- Clinical Trial Center North, Hamburg, Germany